CLINICAL TRIAL: NCT00852371
Title: IPT in Schoolchildren: Comparison of the Efficacy, Safety, and Tolerability of Antimalarial Regimens in Uganda
Brief Title: Intermittent Preventive Treatment of Malaria in Schoolchildren
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Uganda Malaria Surveillance Project (Other); Ministry of Health, Uganda (Other Government)
Responsible Party: Principal Investigator, Brian Greenwood, Professor, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: ITCRVG49; LSHTM Ethics 5197 (Other: London School of Hygiene and Tropical Medicine)
Record Dates: First submitted 2008-02-07; First posted 2009-02-27 (Estimated); Results first posted 2024-03-21 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Malaria; Intermittent Preventive Treatment
Keywords: Malaria; Intermittent preventive treatment; Efficacy; Safety; Tolerability; Schoolchildren; Uganda
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination; Amodiaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Combination of Amodiaquine +sulfadoxine-pyrimethamine (Active Comparator): Combination of Amodiaquine (Camoquin, Parke-Davis, 200 mg tablets, 10 mg/kg on days 0 and 1, and 5 mg/kg on day 2) + sulfadoxine-pyrimethamine (Fansidar, Roche, 500 mg/25 mg tablets, 25 mg/kg sulfadoxine and 1.25 mg/kg pyrimethamine per treatment as a single dose) given as oral tablets
  Interventions: Drug: amodiaquine + sulfadoxine-pyrimethamine
- Dihydroartemisinin-piperaquine (Active Comparator): Dihydroartemisinin-piperaquine (Duocotexin, Holley Pharm, 40 mg dihydroartemisinin/320 mg piperaquine tablets targeting a total dose of 6.4 and 51.2 mg/kg of dihydroartemisinin and piperaquine, respectively, given in 3 equally divided daily doses to the nearest ¼ tablet)
  Interventions: Drug: dihydroartemisinin-piperaquine
- Placebo (Placebo Comparator): Placebo (had no active ingredients, produced by Cosmos Limited, Nairobi, Kenya)
  Interventions: Other: Placebo
- Sulfadoxine-pyrimethamine alone (Active Comparator): sulfadoxine-pyrimethamine (Fansidar, Roche, 500 mg/25 mg tablets, 25 mg/kg sulfadoxine and 1.25 mg/kg pyrimethamine per treatment as a single dose) given as oral tablets
  Interventions: Drug: sulfadoxine-pyrimethamine

INTERVENTIONS:
Drug: sulfadoxine-pyrimethamine — 25 mg/kg po once on day 0
  Other Names: Fansidar, Roche
  Arms: Sulfadoxine-pyrimethamine alone
Drug: amodiaquine + sulfadoxine-pyrimethamine — Amodiaquine: 10 mg/kg po daily for 3 days (on days 0, 1, 2) SP: 25 mg/kg po once on day 0
  Other Names: Camoquin, Pfizer; Fansidar, Roche
  Arms: Combination of Amodiaquine +sulfadoxine-pyrimethamine
Drug: dihydroartemisinin-piperaquine — 2.1/17.1 mg/kg daily for three days (on days 0, 1, 2)
  Other Names: Duocotexcin, Holley Cotec Pharmaceuticals
  Arms: Dihydroartemisinin-piperaquine
Other: Placebo — dosed as for amodiaquine (10mg/kg po daily on days 1, 2)
  Other Names: No active ingredient
  Arms: Placebo

SUMMARY:
This will be a randomized, single-blinded, placebo-controlled trial to evaluate the efficacy, safety and tolerability of antimalarial regimens in healthy schoolchildren. The primary objective of the study is to compare the efficacy of different combination antimalarial regimens, including amodiaquine + sulfadoxine-pyrimethamine (AQ+SP), dihydroartemisinin-piperaquine (DP), and placebo, to SP for intermittent preventive treatment (IPT) in schoolchildren, as measured by risk of parasitaemia (unadjusted by genotyping) after 42 days of follow-up. This will assess both the efficacy for treatment of asymptomatic infections and the efficacy for prevention of new infections.

DETAILED DESCRIPTION:
The study will be carried out among children aged ≥ 8 to < 14 years (boys) and ≥ 8 to < 12 years (girls) attending primary schools in Tororo district. Schools will be selected using convenience sampling with the assistance of the district and the education sector. The target population includes children attending primary schools in Uganda. The accessible population includes the children attending the participating primary schools in classes 3-7 in Tororo district. Children who meet the selection criteria for participation in the study will be randomized to treatment with one of the four study regimens and will be followed for 42 days. Repeat evaluations will be performed on days 1, 2, 3, 7, 14, 28, and 42 (and any unscheduled day that a student is ill) and will include assessment for the occurrence of adverse events. Treatment efficacy outcomes will be assessed using revised WHO outcome classification criteria. Acceptability of treatment regimens will be assessed using a questionnaire administered to participating students on day 7. The primary outcome measure is risk of parasitaemia (unadjusted by genotyping) after 42 days of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 8 to < 14 years (boys), ≥ 8 to < 12 years (girls)
* Student enrolled at participating school in classes 3-7
* Provision of informed consent from parent or guardian
* Provision of assent by student

Exclusion Criteria:

* Known allergy or history of adverse reaction to study medications
* Onset of menstruation (girls)
* Fever (≥ 37.5°C axillary) or history of fever in the previous 24 hours
* Evidence of severe malaria or danger signs
* Haemoglobin < 7.0 gm/dL
* Parasite density > 10,000/ul

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 780 (Actual)
Dates: Start 2008-02; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah G Staedke, MD, Principal Investigator — London School of Hygiene and Tropical Medicine

REFERENCES:
- [Derived] Nankabirwa J, Cundill B, Clarke S, Kabatereine N, Rosenthal PJ, Dorsey G, Brooker S, Staedke SG. Efficacy, safety, and tolerability of three regimens for prevention of malaria: a randomized, placebo-controlled trial in Ugandan schoolchildren. PLoS One. 2010 Oct 19;5(10):e13438. doi: 10.1371/journal.pone.0013438. PMID 20976051

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
Started | 198 | 200 | 196 | 186
Completed | 196 | 197 | 192 | 184
Not Completed | 2 | 3 | 4 | 2
Not completed — Lost to Follow-up | 2 | 3 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Dihydroartemisinin-piperaquine | Placebo | Sulfadoxine-pyrimethamine Alone | Total
Number analyzed (Participants) | 200 | 198 | 196 | 186 | 780
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.7 (1.93) | 10.3 (1.73) | 10.6 (1.86) | 10.6 (1.85) | 10.6 (1.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 87 | 78 | 70 | 313
  Male | 122 | 111 | 118 | 116 | 467
Bed net use [Count of Participants; unit: Participants] | 56 | 56 | 57 | 47 | 216
Mean hemoglobin [Mean (Standard Deviation); unit: g/dL] | 12.7 (1.33) | 12.4 (1.26) | 12.7 (1.38) | 12.7 (1.31) | 12.6 (1.32)

OUTCOME MEASURES:

1. Primary Outcome: Risk of Parasitaemia (Unadjusted by Genotyping)
Description: Proportion of participants whose thick blood smears that are positive for asexual parasites
Time Frame: after 42 days of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
Number analyzed (Participants) | 198 | 200 | 196 | 186
Participants | 23 | 87 | 164 | 147

2. Secondary Outcome: Risk of Recrudescence (Adjusted by Genotyping) in Participants Who Were Parasitaemic at Enrollment
Description: Proportion of participants whose thick blood smears that are positive with the same asexual parasites at baseline and on the day of failure at genotyping
Time Frame: after 42 days of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
Number analyzed (Participants) | 82 | 103 | 109 | 98
Participants | 2 | 6 | 64 | 50

3. Secondary Outcome: Risk of New Infection (Adjusted by Genotyping) in All Participants
Description: Proportion of participants whose thick blood smears that are positive for new asexual parasites on day of failure at genotyping
Time Frame: after 42 days of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
Number analyzed (Participants) | 93 | 113 | 85 | 88
Participants | 12 | 55 | 64 | 62

4. Secondary Outcome: Risk of Clinical Failure Due to Recrudescence (Adjusted by Genotyping) in Children Who Were Parasitaemic at Enrollment
Description: Proportion of children who were parasitaemia at enrollment, with subsequent fever and a positive thick blood smear for asexual parasites on the day of failure during follow-up
Time Frame: Over 42 days of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
Number analyzed (Participants) | 103 | 82 | 109 | 98
Participants | 2 | 6 | 64 | 50

5. Secondary Outcome: Mean Change in Haemoglobin
Description: Haemoglobin measured in g/dL; Mean change in haemoglobin calculated as the difference in mean haemoglobin (g/dL) on Day 42 - Day 0, in children treated with the different antimalarial regimens
Time Frame: Between day 0 to day 42
Measure: Mean (95% Confidence Interval); unit: g/dL
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
Number analyzed (Participants) | 198 | 200 | 196 | 186
g/dL | 0.34 [0.15 to 0.53] | 0.37 [0.18 to 0.56] | 0.24 [0.05 to 0.44] | 0.18 [0.02 to 0.38]

6. Secondary Outcome: Risk of Serious Adverse Events
Description: Any untoward medical occurrence in a participant taking study medication after 14 and 42 days of follow up leading to death, disability, hospitalization or extended hospitalization
Time Frame: over 42 days of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
Number analyzed (Participants) | 198 | 200 | 196 | 186
Participants | 117 | 122 | 125 | 114

7. Secondary Outcome: Acceptability of IPT Regimens
Description: Perceived willingness to take study medication as routine preventive treatment
Time Frame: on day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
Number analyzed (Participants) | 198 | 199 | 195 | 186
Participants | 55 | 67 | 20 | 23

8. Secondary Outcome: Risk of Clinical Failure Due to Recrudescence (Adjusted by Genotyping) in Children Who Were Parasitaemic at Enrollment
Description: as for outcome 4
Time Frame: after 42 days of follow-up
Population: Risk of recrudescence in children with parasites on day 0 (n=392). The risk of recrudescence was estimated using Kaplan-Meier survival techniques with corresponding 95% confidence intervals (CI) calculated using Greenwood variance estimates.
Measure: Count of Participants; unit: Participants
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
Number analyzed (Participants) | 103 | 82 | 109 | 98
Participants | 2 | 6 | 64 | 50

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Dihydroartemisinin-piperaquine | Combination of Amodiaquine +Sulfadoxine-pyrimethamine | Placebo | Sulfadoxine-pyrimethamine Alone
All-Cause Mortality (participants affected / at risk) | 0/198 | 0/200 | 0/196 | 0/186
Serious Adverse Events (participants affected / at risk) | 0/198 | 0/200 | 0/196 | 0/186
Other Adverse Events (participants affected / at risk) | 117/198 | 122/200 | 124/196 | 114/186
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dihydroartemisinin-piperaquine (N=198) | Combination of Amodiaquine +Sulfadoxine-pyrimethamine (N=200) | Placebo (N=196) | Sulfadoxine-pyrimethamine Alone (N=186)
Fever (Infections and infestations) | 6 (6) | 7 (7) | 16 (16) | 10 (10)
Headache (Infections and infestations) | 49 (49) | 53 (53) | 50 (50) | 40 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 54 (54) | 35 (35) | 34 (34) | 32 (32)
Nausea (Gastrointestinal disorders) | 14 (14) | 27 (27) | 24 (24) | 32 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No